CLINICAL TRIAL: NCT05585814
Title: CapeOX Combined With Bevacizumab Plus Pembrolizumab as Neoadjuvant Therapy for Microsatellite Stable Locally Advanced Rectal Cancer (COBP)
Brief Title: CapeOX Combined With Bevacizumab Plus Anti-PD1 Antibody as Neoadjuvant Therapy for Microsatellite Stable Locally Advanced Rectal Cancer
Acronym: COBP
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZHOUHAIYANG
Record Dates: First submitted 2022-10-09; First posted 2022-10-19 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Locally Advanced Colorectal Cancer
MeSH Terms: interventions — Capecitabine; Oxaliplatin; Bevacizumab; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab+ Bevacizumab + CapeOx as neoadjuvant treatment for 4 cycles (Experimental): CapeOx: Capecitabine is given orally at 1000mg / m² twice a day from day1-14 every 3 weeks for 4 cycles and Oxaliplatin is given by intravenous infusion at 130mg / m2 on Day 1 every 3 weeks for 4 cycles;
  Bevacizumab：Bevacizumab is given intravenously at 7.5mg/kg on day 1 every 3 weeks for 4 cycles;
  Pembrolizumab：Pembrolizumab is given intravenously at 200 mg on day 1 every 3 weeks for 4 cycles
  Interventions: Drug: Capecitabine; Drug: Oxaliplatin; Drug: Bevacizumab; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Capecitabine — Capecitabine is given orally at 1000mg / m² twice a day from day1-14 every 3 weeks for 3 cycles
Drug: Oxaliplatin — Oxaliplatin is given by intravenous infusion at 130mg / m2 on Day 1 every 3 weeks for 3cycles
Drug: Bevacizumab — Bevacizumab is given intravenously at 7.5mg/kg on day 1 every 3 weeks for 3 cycles
Drug: Pembrolizumab — Pembrolizumab is given intravenously at 200 mg on day 1 every 3 weeks for 3 cycles

SUMMARY:
This prospective, single-arm study aims to investigate the efficacy and safety of pembrolizumab plus bevacizumab and chemotherapy as neoadjuvant treatment in pMMR/MSS locally advanced rectal cancer patients

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed rectal adenocarcinoma with cT3+N+M0
* Immunohistochemistry and/or genetic testing confirmed pMMR/MSS
* Initial diagnosed or recurrent patients will be accepted, patients with recurrence should not have received any treatment include chemotherapy, targeted therapy or immunotherapy within 1 month or radiotherapy within 1 year
* Measurable disease according to the Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 criteria and haven't received any local treatment.
* Eastern Cooperative Oncology Group (ECOG) 0-1.
* Absence of distant metastasis confirmed by CT, MRI or PET/CT
* Adequate hematologic and organ function, defined by protocol-specified laboratory test results, obtained within 7 days before first dose. Absolute neutrophil count ≥1500/mm3, platelet ≥100,000/mm3, Hb ≥10g/dl, serum creatinine ≤1.5 times ULN, creatinine clearance rate ≥50mL/min, ALT and AST ≤2.5 times ULN, INR or aPTT ≤1.5 times ULN (INR ≤2 times ULN and aPTT in normal range for patients who are on prophylactic anticoagulant therapy within 14 days before study treatment), total bilirubin level ≤2 times ULN (within 7 days before study treatment).
* Women of childbearing age should confirm that serum pregnancy test is negative and agree to use effective contraceptive methods during study treatment and the following 60 days.
* Life expectancy> 3 months
* Signed and written informed consent

Exclusion Criteria:

* Previously received anti-PD1 or anti-PDL1 or anti-PDL2 or anti-CTLA4.
* Uncontrolled active bleeding from the primary tumor or intestinal obstruction.
* Contraindications of bevacizumab
* Hypersensitivity to other monoclonal antibodies.
* Any active, known or suspected autoimmune disease.
* Uncontrolled pleural effusion, pericardial effusion, or ascites to a moderate or greater extent.
* History of one of the following diseases: idiopathic pulmonary fibrosis, organized pneumonia (eg. bronchiolitis obliterans), drug-induced pneumonia, idiopathic pneumonia and interstitial pneumonia, or evidence of active pneumonia through enhanced chest CT screening.
* Major surgery within 4 weeks before enrollment and haven't fully recovered from the previous surgery.
* Active bleeding or abnormal coagulation (aPTT >43s or INR >1.5 times ULN), or having a tendency to bleed or receiving thrombolytic or anticoagulant therapy.
* Previously received allogeneic stem cell or parenchymal organ transplantation.
* Any significant clinical or laboratory abnormality that the investigator considers to influence the safety assessment, eg. uncontrolled active infection, uncontrolled diabetes, hypertension that cannot be reduced to normal range with monotherapy, grade II or above peripheral neuropathy, congestive heart failure, heart disease (class II or higher) as defined by the New York College of Cardiology, myocardial infarction within 3 months prior to enrollment, unstable arrhythmias, unstable angina pectinis, chronic kidney disease, abnormal thyroid function and previous or co-existing malignancies.
* History of uncorrected serum electrolyte disturbances such as potassium, calcium and magnesium.
* HIV infection.
* Active hepatitis B or hepatitis C.
* Pregnancy or lactation period, or unwilling to use contraception during the trial.
* With other malignancy within 5 year, except cervical carcinoma in situ, basal or squamous skin cancer, local prostatic carcinoma and ductal carcinoma in situ.
* Use corticosteroids (dose of prednisone or similar drugs> 10mg/day) or other immunosuppressive agents within 14 days before enrollment.
* Patients with active tuberculosis (TB) who are receiving anti-TB treatment or have received anti-TB treatment within 1 year.
* Active infection, or treatment with oral or intravenous antibiotics within the first 2 weeks prior to neoadjuvant therapy, except prophylactic administration.
* Anti-infective vaccine (eg. influenza vaccine, varicella vaccine, etc.) injection within 4 weeks before neoadjuvant therapy.
* Previous participation in other clinical trials within 4 weeks before neoadjuvant therapy.
* Any other disease, metabolic disorder, abnormal physical examination or abnormal laboratory results that may constrain the use of trial drug, or affect the reliability of study results, or lead to high risk of treatment complications, or affect patient compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
R0 resection rate | 15 weeks
  Percentage of patients who achieve R0 resection
Pathological complete response rate | 15 weeks
  Percentage of patients who achieve pathological complete response (pCR) based on local investigator
Tumor regression grade (TRG) | 15 weeks
Objective response rate | 3 years
  Percentage of patients who achieve partial response (PR) or complete response (CR)

SECONDARY OUTCOMES:
Incidence of Treatment-Related Adverse Events | Until 30 days after the last treatment
  Number of adverse events
Surgical complications | Until 90 days after surgery
Quality of life score (QoL score) | Until 30 days after the last treatment
  Assessment of life quality based on EORTC QLQ-C30
Event free survival | Up to 3 years
  Measure of time from study treatment to disease progression or death
Disease-free survival | Up to 3 years
  Measure of time from the date of surgery to disease relapse or death
One-year or two-year disease-free survival rate | Up to 2 years
  Percentage of patients who achieve disease-free survival lasting for more than one and two years respectively from the date of surgery
One-year or two-year overall survival rate | Up to 2 years
  Percentage of patients who achieve survival for more than one and two years respectively from date of first dose

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Changzheng Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No